CLINICAL TRIAL: NCT02722759
Title: Comparison of Alternative Non-invasive and Invasive Methods of Haemoglobin Measuring With the Gold Standard in Preterm and Term Neonates
Brief Title: Haemoglobin Measurement for Babies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Dr. Eva Wittenmeier:MD, Principal Investigator, Johannes Gutenberg University Mainz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Haemoglobin2016
Record Dates: First submitted 2016-03-10; First posted 2016-03-30 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Hemoglobins; Infant; Non-invasive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hemoglobin measurement arm (Other): In this arm hemoglobin measurement is done by four different devices
  * device "Radical-7" for non-invasive measurement of SpHb
  * device "HemoCue" for taking capillary and venous blood for measurement of HcHb
  * device "ABL 800" for measurement of BGAHb
  * device "Siemens ADVIA" for measurement of labHb
  For measurement of haemoglobin by the devices the following interventions have to be done:
  * venous or arterial puncture (routine)
  * capillary puncture
  * placing of the "Radical 7" sensor
  Interventions: Other: hemoglobin measurement

INTERVENTIONS:
Other: hemoglobin measurement

SUMMARY:
In this prospective study different methods of haemoglobin measurement in term and preterm neonates are compared with the gold standard. Non-invasive haemoglobin measurement with the Radical-7® (SpHb, Masimo®), point-of-care haemoglobin-measurement (HcHb, HemoCue@, Radiometer), blood-gas-analysis (BGAHb,ABL800®, Radiometer) are compared with haemoglobin measurement by an automated hematology analyzer (labHb, Siemens Advia®).

DETAILED DESCRIPTION:
Neonates admitted to neonatal intensive care unit or to a normal neonatal ward are enrolled in the study, if parents have given their written informed consent. Non-invasive SpHb measurements are recorded prior to routine venous sampling. Routine venous sampling includes labHb and BGAHb. Additionally HcHb is taken from the routine venous sampling (HcHbart/ven) and from an additionally capillary puncture of earlobe or heel (HcHbcap). Every neonate can participate in two measurements.

ELIGIBILITY:
gender both

age limits minimum age 3 days of life maximum age 44 postmenstrual weeks

accepts no healthy volunteers

Inclusion Criteria:

written informed consent of the parents

-

Exclusion Criteria:

* allergy against sensor patch
* medical or psychological factors that inhibit a correct finazilation of the study

Ages: 3 Days to 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
accuracy of different methods (SpHb, HcHb,BGAHb) of haemoglobin measurement compared with the gold standard labHb | through study completion, an average of 3 months
  accuracy is assessed by Bland-Altman-method of comparison, by Root mean square error and by out of range

SECONDARY OUTCOMES:
handling of the SpHb-device | through study completion, an average of 3 months
  measurement of how often the Radical-7 has to be replaced and of the time until a stable Signal appears
influence of weight and gender on accuracy of SpHb | through study completion, an average of 3 months
  correlation of PI with the accuracy of SpHb
influence of PI (perfusion index) on accuracy of SpHb | through study completion, an average of 3 months
  correlation of PI with the accuracy of SpHb
influence of concentration of HbF on accuracy of SpHb,BGAHb, HcHb | through study completion, an average of 3 months
  correlation of concentration of HbF with the accuracy of SpHb
influence of concentration of Hb on accuracy of SpHb,BGAHb, HcHb | through study completion, an average of 3 months
  correlation of concentration of Hb with the accuracy of SpHb
agreement of concentration of HbF of BGAHb with HbF of labHb | through study completion, an average of 3 months
  accuracy is assessed by Bland-Altman-method of comparison

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Eva Wittenmeier, Mainz, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wittenmeier E, Lesmeister L, Pirlich N, Dette F, Schmidtmann I, Mildenberger E. Assessment of haemoglobin measurement by several methods - blood gas analyser, capillary and venous HemoCue(R) , non-invasive spectrophotometry and laboratory assay - in term and preterm infants. Anaesthesia. 2019 Feb;74(2):197-202. doi: 10.1111/anae.14481. Epub 2018 Nov 14. PMID 30427065